CLINICAL TRIAL: NCT05294588
Title: Division of Microbiology and Infectious Diseases, (DMID) 21-0018: Efficacy of Immunization With 4C-MenB in Preventing Experimental Urethral Infection With Neisseria Gonorrhoeae
Brief Title: Efficacy of Immunization With 4C-MenB in Preventing Experimental Urethral Infection With Neisseria Gonorrhoeae
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: University of North Carolina, Chapel Hill (Other)
Collaborators: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: 21-0498; DMID 21-0018 (Other: University of North Carolina at Chapel Hill); U01AI162457-01 (NIH)
Record Dates: First submitted 2022-03-15; First posted 2022-03-24 (Actual); Last update posted 2025-03-19 (Actual); Status verified 2025-03

CONDITIONS: Gonorrhea Male
Keywords: 4CMenB; Bexsero; vaccine; controlled human infection model; Neisseria gonorrhoeae
MeSH Terms: interventions — Cefixime; Ceftriaxone; Ciprofloxacin; 4CMenB vaccine; Influenza Vaccines; FluLaval

STUDY DESIGN:
Intervention Model Description: The study intervention is vaccination with two doses of BEXSERO™and with two commercially available FDA-approved vaccines that do not have relevance to Neisseria gonorrhoeae: quadrivalent influenza (FLULAVAL™) and tetanus/diphtheria (TDVAX™). At enrollment, participants are randomized in a 1:1 ratio to the control vaccine arm or the experimental vaccine arm. Participants assigned to the control arm of the study receive immunization with control vaccinations prior to Neisseria gonorrhoeae challenge and with BEXSERO™after Neisseria gonorrhoeae challenge. Participants assigned to the experimental arm of the study receive immunization with BEXSERO™ prior to Neisseria gonorrhoeae challenge and with after control vaccinations Neisseria gonorrhoeae challenge.
Who Masked: Participant, Care Provider, Investigator
Masking Description: Participants and laboratory and clinical staff conducting Ng challenge and assessment of infection and immune responses will be blinded to study arm assignment. Randomization group assignments will be maintained throughout the study.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Experimental arm (Experimental): All participants receive two immunizations prior to the bacterial challenge phase and two immunizations after the challenge phase. Individuals assigned to the experimental arm receive the recommended two doses of BEXSERO™ prior to bacterial challenge and control vaccines (FLULAVAL™ and TDVAX™) in the post-challenge vaccination phase.
  For bacterial challenge, all participants receive a suspension containing 10^6 colony-forming units of N. gonorrhoeae strain FA1090 delivered to the anterior urethra. Participants receive 100% effective antibiotic treatment for N. gonorrhoeae strain FA1090 infection when (1) requested by the participant regardless of signs, symptoms or positive cultures, (2) urethral discharge is observed by the examining clinician or reported by the participant, or (3) 10 days afterurethral inoculation with bacterial product, regardless of infection status.
  Interventions: Drug: Cefixime; Drug: Ceftriaxone; Drug: Ciprofloxacin; Biological: Neisseria gonorrhoeae strain FA1090; Biological: Meningococcal Group B Vaccine; Biological: Influenza Vaccine; Biological: Tetanus-diptheria Vaccine
- Control arm (Other): All participants receive two immunizations prior to the bacterial challenge phase and two immunizations after the challenge phase. Individuals assigned to the control arm receive control vaccines that have no relevance to N. gonorrhoeae infection (FLULAVAL™ and TDVAX™) prior to bacterial challenge and then receive two doses of BEXSERO™ in the post-challenge vaccination phase.
  For bacterial challenge, all participants receive a suspension containing 10^6 colony-forming units of N. gonorrhoeae strain FA1090 delivered to the anterior urethra. Participants receive 100% effective antibiotic treatment for N. gonorrhoeae strain FA1090 infection when (1) requested by the participant regardless of signs, symptoms or positive cultures, (2) urethral discharge is observed by the examining clinician or reported by the participant, or (3) 10 days afterurethral inoculation with bacterial product, regardless of infection status.
  Interventions: Drug: Cefixime; Drug: Ceftriaxone; Drug: Ciprofloxacin; Biological: Neisseria gonorrhoeae strain FA1090; Biological: Meningococcal Group B Vaccine; Biological: Influenza Vaccine; Biological: Tetanus-diptheria Vaccine

INTERVENTIONS:
Drug: Cefixime — Mandatory rescue therapy consisting of cefixime 400 mg orally in a single dose: on patient request, at the onset of clinically apparent urethritis or on the 10th study day after inoculation.
Drug: Ceftriaxone — Mandatory rescue therapy consisting of ceftriaxone 250 mg intramuscularly in a single dose: on patient request, at the onset of clinically apparent urethritis or on the 10th study day after inoculation.
Drug: Ciprofloxacin — Mandatory antibiotic treatment failure therapy: Ciprofloxacin 500 mg orally in a single dose: if the subject has a positive N. gonorrhoeae test within 1 week post initial antibiotic treatment
Biological: Neisseria gonorrhoeae strain FA1090 — 0.4 mL of a suspension containing 10^5 - 10^6 CFU of Neisseria gonorrhoeae, in phosphate-buffered saline, delivered to the anterior urethra through a No.8 pediatric French catheter.
Biological: Meningococcal Group B Vaccine — All participants will receive 2 doses of the 4CMenB vaccine, 0.5 mL intramuscularly
  Other Names: Bexsero; 4-component Neisseria meningitidis group B vaccine; 4CMenB
Biological: Influenza Vaccine — All participants will receive the quadrivalent influenza vaccine, 0.5 mL intramuscularly.
  Other Names: Flulaval
Biological: Tetanus-diptheria Vaccine — All participants will receive the Td vaccine, 0.5 mL intramuscularly.
  Other Names: TDVAX

SUMMARY:
This is a double-blind randomized controlled trial to test whether the group B meningitis vaccine 4 component Neisseria meningitidis serogroup B vaccine (BEXSEROTM) (4C-MenB), trade name Bexsero™), currently approved for use by the United States Food and Drug Administration (FDA) and recommended by the Centers for Disease Control and Prevention (CDC) for protection from Neisseria meningitidis infections, also protects from Neisseria gonorrhoeae infection using controlled human experimental infection to test protection. The information the investigator learn by doing this study may also help to develop a vaccine that protects individuals from having gonorrhea infection.

The study population will consist of male participants > 18 and < 36 years old, living in central North Carolina, in general good health without a history of 4C-MenB vaccination. Approximately 120-140 participants will be enrolled.

Participants will receive 2 doses of vaccine (2 doses of 4C-MenB or 2 comparator vaccines- seasonal influenza and tetanus/diptheria booster) as intramuscular injections, and then one intraurethral challenge with Neisseria gonorrhoeae. Following the challenge, participants will cross-over and receive two doses of vaccines not received prior to challenge (2 doses of 4CMenB or the 2 comparator vaccines- seasonal influenza and tetanus/diptheria booster) All participants receive all vaccinations by the end of the study and all vaccines used in this study are licensed and FDA-approved.

DETAILED DESCRIPTION:
The study is a single-site, double-blind randomized controlled trial to test whether vaccination with 4C-MenB, BEXSERO™ (approved for protection against invasive disease with group B Neisseria meningitidis), according to the FDA-approved schedule , provides protection from urethral infection with Neisseria gonorrhoeae in the controlled human male gonococcal infection model. The study will be conducted in 3 phases: 1) initial vaccination phase, 2) Neisseria gonorrhoeae challenge phase, and 3) post-challenge vaccination phase.

The study intervention is vaccination with two doses of BEXSERO™ and two commercially available FDA-approved vaccines that do not have relevance to Neisseria gonorrhoeae: quadrivalent influenza (FLULAVAL™) and tetanus/diphtheria (TDVAX™). At enrollment, participants are randomized in a 1:1 ratio to the control vaccine arm or the experimental vaccine arm. All participants receive two immunizations prior to the bacterial challenge phase and two immunizations in the post-challenge phase. Individuals assigned to the experimental arm receive two doses of BEXSERO™ prior to Neisseria gonorrhoeae challenge and control vaccines in the post-challenge vaccination phase. Participants assigned to the control arm receive FLULAVAL™ and TDVAX™ prior to challenge and BEXSERO™ in the post-challenge vaccination phase. Primary and secondary outcomes are determined following bacterial challenge. This study design provides clinical equipoise, because all participants receive the known benefits associated with administration of BEXSERO™ for protection against meningococcal disease.

For bacterial challenge, all participants receive a suspension containing 10^6 colony-forming units of Neisseria gonorrhoeae strain FA1090 delivered to the anterior urethra. This dose has been shown to produce symptomatic gonococcal urethritis in 80-90% of unvaccinated, exposed participants within 5 days after bacterial inoculation. Participants are followed with daily visits to assess for development of urethritis and presence of Neisseria gonorrhoeae in their urine. Participants receive 100% effective antibiotic treatment when (1) requested by the participant regardless of signs, symptoms or positive cultures, (2) urethral discharge is observed by the examining clinician or reported by the participant, or (3) 10 days after urethral inoculation with bacterial product, regardless of infection status.

ELIGIBILITY:
Inclusion Criteria:

Participants must meet all the inclusion criteria to participate in the study.

* Assigned male at birth and now ≥ 18 and < 36 years old
* No history of prior Neisseria meningitidis serogroup B (MenB) vaccination
* Able and willing to be located easily by providing street address and telephone number (land line and/or cell phone number)
* Willingness to provide written informed consent
* Informed consent obtained and signed
* Able and willing to attend all study visits
* Able and willing to abstain from all sexual activity involving contact with the participant's penis, urine, or semen and a person other than the participant during experimental gonococcal infection phase until the follow-up test for gonorrhea is negative
* Able and willing to abstain from scheduled immunizations other than those provided through the study, between enrollment and completion of Ng challenge.
* No clinically significant abnormalities on physical exam
* Urinalysis: leukocyte esterase and WBC values within normal limits
* 50% complement hemolytic activity (CH50) within normal limits (WNL)
* Negative HIV and syphilis test results at the screening visit
* Denies history of bleeding diathesis
* Denies history of seizures (due to reports of seizures with ciprofloxacin), history of childhood febrile seizure acceptable
* Denies history of cancer, except basal cell carcinoma of the skin >5 years ago
* Denies current drug abuse that would interfere with study activities
* Denies history of penile, urethral, prostate, testis and associated structures surgery (varicocele repair, vasectomy, and vasectomy repair are acceptable if greater than 1 year prior to enrollment)

Exclusion Criteria:

Participants meeting any of the exclusion criteria at initial screening and screening prior to Ng challenge will be excluded from study participation. If the results of Complete blood count (CBC), serum alanine transaminase (ALT), serum creatinine, or urinalysis obtained at initial screening are outside acceptable limits, and the clinician judges the deviation unlikely to be clinically relevant, one-time repeat screening is permitted. Acceptable laboratory values are presented in Appendix B.15

* Student or employee under the direct supervision of any of the study investigators
* Any known immunodeficiencies, including complement deficiency, antibody deficiency, chronic granulomatous disease or HIV infection
* A history of prior confirmed N. meningitidis infection
* Hemophilia or other bleeding diatheses.
* Autoimmune disorders; mild autoimmune disorders, such as eczema, are not exclusionary and will be determined by the study physician.
* Unstable psychiatric condition (defined as receiving either <3 months of the same medication (and dose) or a decompensating event during the previous 3 months) or psychiatric condition that, in the opinion of the investigator, will compromise the participant's ability to comply with protocol requirements
* Known anatomic abnormality of the urethra or urethral meatus (granular hypospadias is not exclusionary if the study physician believes that the urethral location will not interfere with inoculation catheter insertion)
* Any immunization in 28 days prior to enrollment
* Self-reported treatment for cancer within the past year
* Receipt of anticoagulants (aspirin or nonsteroidal anti-inflammatory drugs (NSAIDS) are acceptable) within 14 days prior to study entry.
* Use of any systemic immunomodulatory treatment, systemic corticosteroids, (inhaled and topical corticosteroids acceptable), investigational products, interleukins, interferons, growth factors, or intravenous immunoglobulin (IVIG) within 45 days prior to study entry.
* Have donated blood or blood products within 28 days before study vaccination, plan to donate blood at any time during the study and up to 28 days after the last blood draw.
* Allergy to penicillin, cephalosporins or ciprofloxacin or to lidocaine or any component of 4C-MenB vaccine or control vaccines (flu, Influenza vaccine (FLULAVALTM) and Td, TDVAXTM), including latex (confirmed delayed contact hypersensitivity to latex is not exclusionary)
* Treatment with medications that are contraindicated with cefixime, ceftriaxone or ciprofloxacin and that cannot be withheld for the single doses given in this study
* Serum creatinine level > 1.1X upper limit of normal (ULN) and deemed clinically significant by the study physician
* Serum ALT level > 1.25X ULN and deemed clinically significant by the study physician
* WBC count < 2.5 or > 15.0 x109/L and deemed clinically significant by the study physician
* Absolute neutrophil count (ANC) < 1.0 x 109/L and deemed clinically significant by the study physician
* Hemoglobin level < 11.0 g/dL or above ULN and deemed clinically significant by the study physician
* Urinalysis: Qualitative protein level ≥ 1+ or Red blood cell (RBC) count≥ 6/hpf
* Any condition in the opinion of the investigator that would interfere with the proper conduct of the trial.

Medications not permitted with cefixime or ceftriaxone:

Warfarin Probenecid Aspirin Diuretics such as furosemide Aminoglycoside antibiotics Chloramphenicol

Medications not permitted with ciprofloxacin:

Tizanidine Theophylline Warfarin Glyburide Cyclosporine Probenecid Phenytoin Methotrexate Antacids, multivitamins, and other dietary supplements containing magnesium, calcium, aluminum, iron or zinc Caffeine-containing medications Sucralfate or didanosine chewable or buffered tablets

Ages: 18 Years to 35 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Participants assigned male sex at birth any race or ethnicity
Enrollment: 140 (Estimated)
Dates: Start 2022-04-18 (Actual); Primary Completion 2028-02 (Estimated); Study Completion 2028-02 (Estimated)

PRIMARY OUTCOMES:
Infectivity of N. gonorrhoeae inoculum | between 1 and 10 days after N. gonorrhoeae inoculation (between study day 58 and study day 123)
  Infectivity is defined as the proportion of participants positive for N. gonorrhoeae by N. gonorrhoeae Nucleic acid amplification tests (NAAT) or urine culture or swab culture on the post-inoculation antibiotic treatment day in each study group (control and experimental).

SECONDARY OUTCOMES:
Proportion of participants that develop macroscopic urethritis | between 1 and 10 days after N. gonorrhoeae inoculation (between study day 58 and study day 123)
  The proportion of participants with protocol defined macroscopic urethritis on the post-inoculation antibiotic treatment day in each study group (control and experimental).
Proportion of participants that develop symptomatic microscopic urethritis | between 1 and 10 days after N. gonorrhoeae inoculation (between study day 58 and study day 123)
  The proportion of participants with protocol defined symptomatic microscopic urethritis on the post-inoculation antibiotic treatment day in each study group (control and experimental).
Time to develop macroscopic urethritis | between 1 and 10 days after N. gonorrhoeae inoculation (between study day 58 and study day 123)
  The time to develop macroscopic urethritis is defined as the number of days after urethral inoculation with N. gonorrhoeae to the day that protocol defined macroscopic urethritis triggers antibiotic treatment will determined for each study group (control and experimental)

CONTACTS AND LOCATIONS:
Overall Officials: Joseph A Duncan, MD, PhD, Principal Investigator — University of North Carolina, Chapel Hill
Locations (1):
- Clinical and Translational Research Center (CTRC) at University of North Carolina (UNC) Hospitals and/or at UNC Global Clinical Research North, Chapel Hill, North Carolina, United States

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual data that supports the results will be shared beginning 12 to 24 months following publication provided the investigator/researcher who proposes to use the data has approval from an Institutional Review Board (IRB), Independent Ethics Committee (IEC), or Research Ethics Board (REB), as applicable, and executes a data use/sharing agreement with UNC.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: 12-24 months after completion
Access Criteria: Investigator/researcher who proposes to use the data IRB, IEC, or REB approval and an executed data use/sharing agreement with UNC.

REFERENCES:
- [Derived] Firth C, Emary K, Stuart A, Browne R, Williamson M, Francis E, Vanderslott S, Hodgson SH. Acceptability of the gonorrhoea human challenge model to accelerate vaccine development in UK men. Vaccine. 2025 Apr 30;54:127013. doi: 10.1016/j.vaccine.2025.127013. Epub 2025 Mar 13. PMID 40086037